CLINICAL TRIAL: NCT05401396
Title: Swimming Immediately After Having a Meal: a Randomized Controlled Study
Brief Title: Swimming Immediately After Having a Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Sehriban Harmankaya, Principal Investigator, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 052022
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Sadness

STUDY DESIGN:
Intervention Model Description: Each participant will on the first day of the trial be randomized either to swim in a pool immediately after lunch or to wait 30 minutes before swimming. The participants will do the opposite on the second day of the trial. The randomization will be done by throwing a dice.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swimming immediately after eating (Experimental): Two arms but all participants are performing both the intervention and the comparison.
  Interventions: Other: Swimming immediately after eating
- Swimming 30 minutes after eating (No Intervention): Two arms but all participants are performing both the intervention and the comparison.

INTERVENTIONS:
Other: Swimming immediately after eating — After having the last bite of lunch, the participants will swim in the pool with a specific distance.
  Arms: Swimming immediately after eating

SUMMARY:
Many believe that it is unsafe to swim immediately after having a meal and that it is preferable to wait at least 30 minutes. The fear is that swimming can cause stomach cramps and muscle cramps with discomfort and potentially drowning.

With this randomized controlled trial, the aim was to investigate whether there was any hold in this belief and what could potentially happen by swimming with the stomach full immediately after a meal.

DETAILED DESCRIPTION:
All volunteers will be adults. Participants will receive both oral and written information about the trial prior to giving consent for participation.

Participants will act as their own control over two days. On the first day, participants will be randomized to either swim immediately after they have eaten their usual lunch or 30 minutes after the last bite. They will do the opposite on the second day. The randomization will be done by throwing a dice.

Prior to swimming, participants will fill out the following:

* Visual analogue scale (VAS) about their well-being
* Questionnaire about their mood state

After swimming, participants will fill out the following:

* Visual analogue scale (VAS) about their well-being
* Questionnaire about their mood state
* Adverse events

Prior to swimming and afterwards, the participants' blood pressure, pulse, and blood oxygen levels will be measured.

Sample size: Convenience sample.

Withdrawal and dropout criteria: All participants will be informed that they can withdraw their consent at any point during the trial without having to explain any reasons.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Healthy volunteers
* Otherwise, no restriction since each participant acts as their own control

Exclusion Criteria:

* Smoking one hour prior to swimming
* Participants who cannot swim

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-05-28 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of mortality | During swimming
  Any adverse events leading to death

SECONDARY OUTCOMES:
Swimming time | During swimming
  Measured by seconds
Discomfort | During the actual swimming and immediately after swimming is completed
  Self-reported assessment of discomfort on a visual analogue scale. Minimum: 0. To Maximum: 100mm. Ranging from no discomfort to the worse imaginable discomfort.
Mood changes | Baseline and immediately after swimming
  Measured by the Profile of mood states. A five-point scale indicating the level of affection. Minimum: 1. To Maximum: 5.
Number of patients with any adverse events | During and immediately after swimming is completed
  Any adverse events other than already mentioned outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Perioperative Optimisation, Department of Surgery, Herlev og Gentofte Hospital, University of Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No